CLINICAL TRIAL: NCT01882686
Title: Efficacy of a Classification Based 'Cognitive Functional Therapy' in Nurses With Non Specific Chronic Low Back Pain - a Series of Case-controls
Brief Title: Efficacy of a Classification Based 'Cognitive Functional Therapy' in Nurses With Non Specific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: European Social Fund (Other)
Responsible Party: Principal Investigator, Prof. dr. Wim Dankaerts, Prof. dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S54606
Record Dates: First submitted 2013-06-12; First posted 2013-06-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Chronic Low Back Pain
Keywords: Pain; Back Pain; Low Back Pain; Chronic Low Back Pain; Cognitive Functional Therapy; Intervention; Subclassification; Multidimensional
MeSH Terms: conditions — Pain; Back Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Classification Based Cognitive Functional Therapy (Experimental)
  Interventions: Other: Classification Based Cognitive Functional Therapy

INTERVENTIONS:
Other: Classification Based Cognitive Functional Therapy — A novel multidimensional classification system has been developed incorporating the biopsychosocial model, which subgroups patients based on their presentation. This subclassification is the base for matched interventions directed at the maladaptive cognitive, physical and lifestyle behaviours associated with the disorder. The intervention is called 'cognitive functional therapy' as it directly challenges these behaviours in a functionally specific and graduated manner.
  Other Names: cognitive functional therapy

SUMMARY:
A series of case-studies to explore the efficacy of classification based cognitive functional physiotherapy according to the classification system proposed by Peter O'Sullivan in specific nursing population with non specific chronic low back pain.

The investigators hypothesis was that treatment targeting the mechanisms behind the problem from a multidimensional perspective would be effective to reduce pain, disability and sick-leave.

DETAILED DESCRIPTION:
Low back pain (LBP) is a common, recalcitrant and costly health problem, which limits patients' daily activities. In 85% of the cases, LBP is classified as 'non-specific', which means there is no clear underlying patho-anatomical/radiological abnormality. This subgroup often gives rise to a chronic fluctuating problem. Although most cases of LBP resolve within 8 to 12 weeks, it may become chronic in up to 15% of patients. LBP constitutes an enormous and growing medical and socio-economical problem for the modern society. Nursing has been identified amongst the top professions at risk for occupational LBP, with lifetime prevalence between 66%-82%. The impact of LBP for nurses includes time off work, increased risk of chronicity, associated personal and economic costs and reduced nursing workforce efficiency.

Non Specific Chronic Low Back Pain (NSCLBP) is widely viewed as a multifactorial biopsychosocial pain syndrome. It has been proposed by several authors that NSCLBP represents a vicious cycle associated with different combinations of maladaptive; cognitive (negative beliefs, fear avoidance behaviours, catastrophising, depression, stress, lack of pacing and coping), physical (pain provocative postures, movement patterns and pain behaviours) and lifestyle (inactivity, rest) behaviours that act to promote pain and disability. However a recent systematic review suggests that this change in paradigm and the investigators new understanding of NSCLBP has not resulted in clinical trials utilizing multidimensional classification systems or targeted interventions based on the underlying mechanisms. In line with this paradigm shift a novel multidimensional classification system has been developed incorporating the biopsychosocial model, which subgroups patients based on their underlying pain mechanism. Enabling a classification based interventions targetting the maladaptive cognitive, physical and lifestyle behaviours associated with the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Low Back Pain (LBP) with/without referred pain in buttock/thigh for > 3 months, including the four weeks prior to testing
* LBP is primarily localised from T12 to gluteal folds
* mechanical provocation of LBP with postures, movement and activities
* average pain intensity in the past week Numerical Rating Scale (NRS) >/= 1/10
* Disability (ODI) >/=2%
* willingness to sign the informed consent

Exclusion Criteria:

* specific spinal pathology
* presence of red flags
* previous lumbar spinal surgery
* pregnancy
* diagnosed psychiatric disorder - somatisation
* radicular pain with positive neural tissue provocation test
* widespread non-specific pain disorder (no primary LBP focus)
* specific diagnoses: active rheumatologic disease, progressive neurological disease, serious cardiac or other internal medical condition, malignant basic diseases, acute traumas, infections, or acute vascular catastrophes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain | 3, 6, 9 and 12 months
  Pain was assessed using a numerical pain rating scale (NPRS) ranging from 0 (no pain) to 10 (worst imaginable pain)
Change from baseline in disability | 3, 6, 9 months, 1 and 3 year
  Disability was measured using the Oswestry Disability Index (ODI)

SECONDARY OUTCOMES:
Change from baseline in Beliefs about LBP | 3, 6, 9 and 12 months
  Back Beliefs Questionnaire (BBQ)
Change from baseline in Chance of long-term disability and failure to return to work | 3, 6, 9 and 12 months
  Tha Acute Low Back Pain Screening Questionnaire (Dutch version of the Ørebro Pain Screening Questionnaire) is a 'yellow flag' screening tool that predicts long-term disability and failure to return to work due to personal and environmental factors.
Change from baseline in Physical activity | 3, 6, 9 and 12 months
  Baecke questionnaire
Change from baseline in Sleep problems | 3, 6, 9 and 12 months
  Insomnia Severity Index (ISI)
Change from baseline in Depression, anxiety and stress | 3, 6, 9 and 12 months
  Depression Anxiety and Stress scale (DASS-21)
Change from baseline in Self-efficacy, coping | 3, 6, 9 and 12 months
  Pain Self-Efficacy Questionnaire (PSEQ)
Change from baseline in Fear-avoidance / kinesiophobia | 3, 6, 9 and 12 months
  Tampa Scale of Kinesiophobia (TSK-17)
Change from baseline in Pain catastrophizing | 3, 6, 9 and 12 months
  Pain Catastrophizing Scale (PCS)
Change from baseline in Psychosocial job aspects | 3, 6, 9 and 12 months
  The Job Content Questionnaire (JCQ) is a tool for psychosocial job assessment.
Change from baseline in Lower Lumbar spine Kinematics | 3, 6, 9 and 12 months
  Lower Lumbar kinematics of the spine were measured with the BodyGuard (sels-instruments nv). This is a remote measuring system.
Patient satisfaction of the intervention | 3, 6, 9 and 12 months
  Patients' Global Impression of Change (PGIC) scale
Change from baseline in Category of risk of poor outcome (persistent disabling symptoms) | 3, 6, 9 and 12 months
  The Start Back Screening Tool is used to screen primary care patients with low back pain for prognostic indicators that are relevant to initial decision making. The tool helps to group patients into 3 categories of risk of poor outcome (persistent disabling symptoms) - low, medium, and high-risk.
Change from baseline in Psychosocial aspects of work | 3, 6, 9 and 12 months
  Psychosocial Aspects of Work Questionnaire (PAWQ)

CONTACTS AND LOCATIONS:
Overall Officials: Wim Dankaerts, Principal Investigator — KU Leuven
Locations (1):
- Lindelo, Lille, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vibe Fersum K, O'Sullivan P, Skouen JS, Smith A, Kvale A. Efficacy of classification-based cognitive functional therapy in patients with non-specific chronic low back pain: a randomized controlled trial. Eur J Pain. 2013 Jul;17(6):916-28. doi: 10.1002/j.1532-2149.2012.00252.x. Epub 2012 Dec 4. PMID 23208945
- [Background] O'Sullivan P. Diagnosis and classification of chronic low back pain disorders: maladaptive movement and motor control impairments as underlying mechanism. Man Ther. 2005 Nov;10(4):242-55. doi: 10.1016/j.math.2005.07.001. Epub 2005 Sep 9. PMID 16154380
- [Background] Dankaerts W, O'Sullivan P. The validity of O'Sullivan's classification system (CS) for a sub-group of NS-CLBP with motor control impairment (MCI): overview of a series of studies and review of the literature. Man Ther. 2011 Feb;16(1):9-14. doi: 10.1016/j.math.2010.10.006. Epub 2010 Nov 20. PMID 21094624
- [Derived] Van Hoof W, O'Sullivan K, Verschueren S, O'Sullivan P, Dankaerts W. Evaluation of Absenteeism, Pain, and Disability in Nurses With Persistent Low Back Pain Following Cognitive Functional Therapy: A Case Series Pilot Study With 3-Year Follow-Up. Phys Ther. 2021 Jan 4;101(1):pzaa164. doi: 10.1093/ptj/pzaa164. PMID 32949123